CLINICAL TRIAL: NCT05806450
Title: Development of a Cognitive-Behavioral Intervention to Improve Infant and Parent Sleep Based on Big Data Analytics
Brief Title: Development of Sleep Intervention for Parent and Child
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sungshin Women's University (Other)
Collaborators: National Research Foundation of Korea (Other)
Responsible Party: Principal Investigator, Sooyeon Suh, Associate professor, Sungshin Women's University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NRF-2021S1A5A2A03061721
Record Dates: First submitted 2023-03-28; First posted 2023-04-10 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Behavioral Insomnia of Childhood
Keywords: pediatric sleep problems; sleep intervention; cognitive behavioral therapy (CBT)
MeSH Terms: interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention condition (Experimental): Structured online intervention consists of three weekly sessions of cognitive therapy and psychoeducation about child sleep
  Interventions: Behavioral: Intervention
- Active control condition (Active Comparator): Psychoeducation about basic sleep structure and sleep hygiene
  Interventions: Other: Active control condition

INTERVENTIONS:
Behavioral: Intervention — Structured online intervention consists of three weekly sessions of cognitive therapy and psychoeducation about child sleep
  Other Names: Sleep Intervention for Mother and BAby (SIMBA)
  Arms: Intervention condition
Other: Active control condition — Psychoeducation about basic sleep structure and sleep hygiene
  Arms: Active control condition

SUMMARY:
This study aims to develop and test the intervention program to help manage parental thoughts in parents with child sleep problems.

DETAILED DESCRIPTION:
Pediatric sleep problems are common and persistent, which result in negative outcomes without appropriate intervention. Behavioral sleep interventions (BSI) are evidence-based sleep training methods for improving pediatric sleep. However, parental factors (e.g., parental dysfunctional beliefs about child sleep) can interfere with the implementation of BSI. For example, being too worried or having misperceptions about infant sleep may interfere with the parent's ability to successfully and persistently implement BSIs. Therefore, parental thoughts and beliefs should be considered as an important target in the context of pediatric sleep interventions. This study aims to develop a cognitive intervention that identifies and targets parental misperceptions about child's sleep, and test the efficacy of the intervention through a randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Child's primary nighttime caregiver (mothers or fathers) of full-term, healthy, singleton, 6 to 24 months old
* Caregiver participants aged between 19 to 65 years
* The caregiver who is a native speaker of Korean (a person who is able to listen, speak, and write in Korean, and does not have any difficulties in understanding the Korean language)
* Residents of South Korea
* Sleep arrangements without restriction for using an auto-videosomnography device: (1) parent-child sleep separately (one should not change the sleep arrangement only for the participation in the study); (2) if parents and child share a bed, the child's own space should be large enough for the videosomnography camera to capture child body solely.
* Be available on devices with the camera (e.g., tablets, personal computers) for the online intervention/session

Exclusion Criteria:

* Child's gestational age before 37 weeks or after 42 weeks
* Children with developmental disability
* Caregiver participant (or partner) who is currently working the night shift or night duty
* Caregiver participant who has a history of sleep disorders besides insomnia
* Caregiver participant who has lifetime bipolar disorder, schizophrenia spectrum, and other psychotic disorders, alcohol, caffeine, or other substance substance-related disorders, neurocognitive disorders, thyroid-related disorders, or epilepsy
* Caregiver participant who is currently experiencing a major depressive disorder, panic disorder (only if ≥ 4 nocturnal panic attacks in the past month), or post-traumatic stress-related problems
* Caregiver participant who is using medications or substances that directly affect sleep
* Caregiver participant who is currently getting cognitive behavioral therapy for insomnia (CBTi)
* Pregnant women

Ages: 6 Months to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 190 (Estimated)
Dates: Start 2023-03-10 (Actual); Primary Completion 2025-06-11 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Parental cognition about child sleep | Changes from baseline to 4 weeks, and 4 weeks and 12 weeks post-intervention
  Parental cognition about child's sleep will be measured by the Parental Understanding and Misperceptions about BAby Sleep-Questionnaire (PUMBA-Q). The score range is 0 to 92. Higher score represents higher levels of maladaptive cognition.
Child sleep diary | Changes from baseline to 4 weeks, and 4 weeks and 12 weeks post-intervention
  Parent-report child's sleep diary will be collected. Sleep parameters include bedtime, wake time, total sleep time, sleep onset latency, wake time after sleep onset, and the number of awakenings. Total sleep time will be used as the main outcome.
Child sleep (objective measurement) | changes from baseline to 4 weeks
  Child sleep will be objectively measured using the videosomnography. Sleep parameters such as bedtime, wake time, total sleep time, sleep onset latency, wake time after sleep onset, number of parental interventions, and number of awakenings are calculated by the algorithm. Total sleep time will be used as the main outcome.

SECONDARY OUTCOMES:
Parental sleep diary | changes from baseline to 4 weeks, and 4 weeks and 12 weeks post-intervention
  Self-report parental sleep diary will be collected. Sleep parameters include bedtime, wake time, total sleep time, sleep onset latency, wake time after sleep onset, and number of awakenings.
Parental sleep (objective measurement) | changes from baseline to 4 weeks
  Parental sleep will be objectively measured by the Fitbit wearable device. Sleep parameters such as bedtime, wake time, and total sleep time are calculated by the algorithm.
Parental insomnia | changes from baseline to 4 weeks, and 4 weeks and 12 weeks post-intervention
  The ISI (Insomnia Severity Index) scale will be used to assess self-reported levels of insomnia severity. Scores range from 0 to 28. Higher scores reflect higher levels of insomnia symptom severity.
Parental sleep disturbance | changes from baseline to 4 weeks, and 4 weeks and 12 weeks post-intervention
  The GSDS (General Sleep Disturbance Scale) scale will be used to assess self-reported levels of general sleep disturbance. Scores range from 0 to 147. Higher scores reflect higher levels of sleep disturbance.
Child sleep environment and parental interaction | changes from baseline to 4 weeks, and 4 weeks and 12 weeks post-intervention
  The Brief Infant Sleep Questionnaire-Revised (BISQ-R) scale will assess child sleep environment such as bedroom environment, sleep routine, and parental behavior around infant sleep.
Anxiety | changes from baseline to 4 weeks, and 4 weeks and 12 weeks post-intervention
  The PROMIS-anxiety scale will be used to assess self-reported levels of anxiety. Scores range from 8 to 40. Higher scores reflect higher levels of anxiety.
Depression | changes from baseline to 4 weeks, and 4 weeks and 12 weeks post-intervention
  The PROMIS-depression scale will be used to assess self-reported levels of depression. Scores range from 8 to 40. Higher scores reflect higher levels of depression.

OTHER OUTCOMES:
Parental cognition about sleep | changes from baseline to 4 weeks, and 4 weeks and 12 weeks post-intervention
  The DBAS-16 (Dysfunctional Beliefs and Attitudes about Sleep-16) scale will be used to assess parental cognition about own sleep. Scores range from 0 to 10. Higher scores reflect more maladaptive cognition.
Marital satisfaction | changes from baseline to 4 weeks, and 4 weeks and 12 weeks post-intervention
  The MSI-B (Marital Satisfaction Index-Brief) scale will be used to assess marital satisfaction. Scores range from 0 to 10. Higher scores reflect worse marital satisfaction.
Circadian rhythm | baseline assessment to identify circadian types that reflect an individual's preferred time of day for activity
  The MEQ (Morningness-Eveningness Questionnaire) scale will be used to assess one's circadian preference. Scores range from 16-86. Higher score means one's circadian preference is more close to morningness.

CONTACTS AND LOCATIONS:
Overall Officials: Sooyeon Suh, PhD, Principal Investigator — Sungshin Women's University
Locations (1):
- Sungshin Women's University, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No